CLINICAL TRIAL: NCT00797706
Title: A Phase I/II Double-Blind, Dose Ranging, Vehicle Controlled, Randomized, Parallel Groups, Safety, Tolerability and Efficacy Study of CHRONSEAL® (5-amino-acid Deleted Recombinant Human Hepatocyte Growth Factor (KP-dHGF)), in Subjects With Venous Leg Ulcers
Brief Title: Phase I/II Dose Ranging CHRONSEAL® Study in Venous Leg Ulcers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kringle Pharma Europe AB (Industry)
Collaborators: Kringle Pharma, Inc. (Industry)
Responsible Party: Prof. Anders Vahlne/CEO, Kringle Pharma Europe AB
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS-201; EudraCT No. 2007-002695-34
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Venous Leg Ulcers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle (Placebo Comparator)
  Interventions: Drug: CHRONSEAL
- Low dose (Experimental)
  Interventions: Drug: CHRONSEAL
- High dose (Experimental)
  Interventions: Drug: CHRONSEAL

INTERVENTIONS:
Drug: CHRONSEAL — Cream (1.4/2.8 g depending on ulcer size) topical administration, every 2nd day at 3 occasions

SUMMARY:
The purpose of this study is to evaluate if the investigational medicinal product CHRONSEAL intended for future treatment of chronic venous leg ulcers is safe and tolerated and if it has an ulcer size reduction effect when administered to individuals suffering from venous leg ulcers.

ELIGIBILITY:
Inclusion criteria (Run-in period):

1. Caucasian male or clinically sterile female subjects
2. 40 years or older.
3. Ankle brachial index of at least 0.6.
4. Written informed consent obtained.
5. Subject legally competent and able to communicate effectively.
6. Subject likely to co-operate.
7. Uncomplicated venous ulcer as by clinical diagnosis.
8. Full skin ulcer.
9. Localisation above the foot and below the knee (wrist and malleoli included)
10. Duration of at least 3 months.
11. Area 3-20 cm2.

Exclusion criteria (Run-in period)

1. Visible signs of infection, black necrosis or discharge in the target ulcer.
2. More than ~20% slough after debridement.
3. Ulcer that by location or extension will either be difficult to follow or to treat according to the protocol.
4. Other known etiology of the target ulcer.
5. Subject having to the discretion of the investigator clinically significant findings on physical examination or vital signs.
6. Concomitant systemic or topical treatment within 14 days prior to start of study medication with antibiotics or antiseptics for treatment of ulcer infection in target ulcer.
7. Concomitant systemic treatment within 14 days prior to start of study medication with immunosuppressives
8. Concomitant topical treatment within 14 days prior to start of study medication with any of the following:

   * NSAIDs, aspirin
   * Growth factors, or other biologically active agents
   * Products containing chlorhexidine, potassium permanganate, iodine or silver
9. Diabetes Mellitus requiring pharmaceutical treatment.
10. Co-morbidity with a life expectancy less than 6 months.
11. Co-morbidity expected to lower compliance.
12. Diagnosed kidney disease
13. Individuals sensitive to any of the study medication components.
14. Subject having received an investigational drug product, or been enrolled in other investigational drug protocols within a period of 30 days prior to receiving the first dose of the study medication.
15. Known abuse of alcohol, drugs or pharmaceuticals.
16. Diagnosis of squamous epithelia carcinoma
17. Diagnoses of a serious psychiatric illness which may influence study participation.

Inclusion criteria (Randomization)

1. Subject likely to co-operate.
2. Ulcer area reduction less than 50% during run-in period.
3. Ulcer area 3-20 cm2.

Exclusion criteria (Randomization)

1.& 2. = Run-in period criteria 1. & 2.

3. Subject having to the discretion of the investigator clinically significant findings on vital signs or laboratory values.

4.-10. = Run-in period criteria 6., 7., 8., 11., 12., 13., & 14

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To investigate safety and local tolerance of CHRONSEAL® cream containing 2 different concentrations of API, applied at 3 occasions every second day in chronic venous leg ulcers compared to vehicle. | From start of treatment to 12 weeks post treatment

SECONDARY OUTCOMES:
To investigate the treatment effect on ulcer area reduction and changes of ulcer condition of CHRONSEAL® cream, containing 2 different concentrations API, applied at 3 occasions every second day in chronic venous leg ulcers compared to vehicle. | From start of treatment to 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hans Olav Høivik, MD, Principal Investigator — Medi 3 Innlandet AS, avd Hamar; Karin Andersson, MD, Principal Investigator — Halland County Council, Department of Dermatology and Infectious diseases, Halmstad, Sweden; Jan Apelqvist, Assoc. Prof., PhD, MD, Study Chair — Department of Endocrinology, University Hospital Malmö,
Locations (16):
- Norway (4):
  - Medi3 Innlandet AS, Department Elverum, Elverum
  - Hudavdelingen Helse, Førde
  - Medi 3 Innlandet AS, Department Hamar, Hamar
  - Colosseumklinikken, Oslo
- Sweden (12):
  - Vårdcentralen Alvesta, Alvesta
  - Danderyds Sjukhus AB, Danderyd
  - Carema Vårdcentral Gubbängen, Enskede
  - Department of Dermatology and Infectious diseases, Halmstad
  - Husläkarna i Kungsbacka, Kungsbacka
  - Department of Dermatology, Lund University hospital, Lund
  - Department of Dermatology, University Hospital MAS, Malmo
  - Gamla Stans Vårdcentral, Stockholm
  - Taptogatans Husläkare, Stockholm
  - Department of Dermatology, Norrlands University hospital, Umeå
  - Department of Medical Sciences, Section of Dermatology and Venereology, Uppsala University hospital, Uppsala
  - Neptunuskliniken, Varberg